CLINICAL TRIAL: NCT02983981
Title: An Open-Label, Observational Study Evaluating Topicort® Topical Spray 0.25% (Desoximetasone) BID in Psoriasis Patients Being Treated With Biologic Agents
Brief Title: Topical Psoriasis Study for Patients Receiving Biologic Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JB-01
Record Dates: First submitted 2016-10-05; First posted 2016-12-06 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental): Topicort topical spray
  Interventions: Drug: Topicort Topical Spray

INTERVENTIONS:
Drug: Topicort Topical Spray — open label Topicort spray

SUMMARY:
A two-phase, single center, study of 20 subjects to assess 4 weeks of add-on therapy of Topicort® BID and 12 weeks BID on two consecutive days a week to patients with ≤5% BSA who are receiving biologic therapy for at least 24 weeks

DETAILED DESCRIPTION:
A two-phase, single center, study of 20 subjects to assess 4 weeks of add-on therapy of Topicort® BID and 12 weeks BID on two consecutive days a week to patients with ≤5% BSA who are receiving biologic therapy for at least 24 weeks.

Adult male and female subjects with moderate to severe chronic plaque psoriasis All patients will receive Topicort® BID for 4 weeks.

After week 4 patients will receive Topicort® BID on two consecutive days a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ≥ 18 years of age.
2. Diagnosis of chronic plaque-type psoriasis.
3. Able to give written informed consent prior to performance of any study related procedures.
4. Treated with a biologic agent for a minimum of 24 weeks at baseline.
5. Plaque-type psoriasis as defined at screening and baseline by BSA ≤ 5%.
6. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options: hormonal contraception; intrauterine device (IUD); tubal ligation; or partner's vasectomy; Male or female condom diaphragm with spermicide, cervical cap with spermicide, or contraceptive sponge with spermicide.
7. Subject must be in general good health (except for psoriasis) as judged by the Investigator, based on medical history, physical examination.

Exclusion Criteria:

1. >5% Body Surface Area
2. Any condition, which would place the subject at unacceptable risk if he/she were to participate in the study.
3. Pregnant or breast feeding, or considering becoming pregnant during the study.
4. Malignancy or history of malignancy, except for:

   1. treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
   2. treated [ie, cured] malignancy with no evidence of recurrence within the previous 5 years.
5. Use of any investigational drug within 4 weeks prior to randomization, or within 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
6. Use of oral systemic medications for the treatment of psoriasis within 4 weeks (includes, but not limited to, oral corticosteroids, methotrexate, acitretin, apremilast and cyclosporine).
7. Patient used other topical therapies to treat within 2 weeks of the Baseline Visit (includes, but not limited to, topical corticosteroids, vitamin D analogs, or retinoids).
8. Patient received UVB phototherapy within 2 weeks of Baseline.
9. Patient received PUVA phototherapy within 4 weeks of Baseline.
10. Patient has a known hypersensitivity to the excipients of Topicort Spray® as stated in the label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Bagel, MD, Principal Investigator — Director

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Topicort Topical Spray: Topicort spray applied BID for 4 weeks followed by BID on 2 consecutive days through week 16
Period: Overall Study
Arm/Group | Topicort Topical Spray
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label: Topicort topical spray
  Topicort Topical Spray: open label Topicort spray applied twice daily for 4 weeks followed by twice daily BID on two consecutive days a week (e.g. Saturday and Sunday) for 12 weeks.
Arm/Group | Open Label
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.33 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Severity
Description: Physician's Global Assessment x Percentage of Body Surface Area (scale scores 0-400 where 0 is best psoriasis 400 is worst possible psoriasis) Body surface area calculated as 1 of patient's palm is 1%.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 20
units on a scale | 4.25 (5.71)

2. Secondary Outcome: Psoriasis Severity
Description: Physician's Global Assessment Scores Scales 0-4 with 0 as no psoriasis and 4 is severe psoriasis
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 20
units on a scale | 1.65 (.89)

3. Secondary Outcome: Psoriasis Severity
Description: Psoriasis severity measured as Body Surface area measured as 1 of patient's palm is equal to 1% body surface area.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Open Label
Number analyzed (Participants) | 20
percentage of BSA | 2.05 (2.28)

4. Secondary Outcome: Dermatology Life Quality Index
Description: calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 20
units on a scale | 3.65 (4.08)

ADVERSE EVENTS:
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=20)
worsening of psoriasis (Skin and subcutaneous tissue disorders) | 2 (2)
erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
sciatic neuralgia (Nervous system disorders) | 1 (1)
cough/congestion (Infections and infestations) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT02983981/Prot_SAP_000.pdf